CLINICAL TRIAL: NCT01738945
Title: Effect of Calcium Channel Blocker on the Serum Fibrobalst Growth Factor-23 (FGF-23) Levels in Type-2 Diabetic Patients With Proteinuria Purpose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mahmut Ilker Yilmaz, Associate Profesoor, Gulhane School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: GATACCBFGF23
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2008-02

CONDITIONS: We Searched for the Effects of Calcium Channel Blocker Amlodipine on the Clinical and Laboratory Parameters of Diabetic Patients With Proteinuria.
MeSH Terms: interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Amlodipine (Other): Amlodipine 10 mg/day for 12 weeks
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — 10 mg/day for 12 weeks

SUMMARY:
In recent years, diabetic nephropathy, which may lead to dialysis treatment, is the most prevalent underlying disease of people in developed countries. A wide range of studies have been carried out, from various points of view, to understand the progress of renal dysfunction in diabetic nephropathy.

Fibroblast growth factor 23 (FGF-23) is a primary regulator of renal phosphate excretion. FGF23 is inversely associated with the GFR, a relationship underlying a fundamental mechanism for maintaining serum phosphate constancy during CKD progression. Such an adaptation may have deleterious trade-offs because, independently of serum phosphate, high FGF23 signals a high risk of death in ESRD patients. Some studies showed that there is relationship between FGF-23 levels and proteinuria in CKD patients.

There is no data about the effects of calcium channel blocker on FGF23 levels in diabetic patients with proteinuria. The aim of this study was to find out whether the beneficial effects of calcium channel blocker in diabetic proteinuria has any relation with the alteration of FGF-23 levels. The investigators searched for the effects of calcium channel blocker amlodipine on the clinical and laboratory parameters of diabetic patients with proteinuria.

The investigators registered the study 'The effect of renin angiotensin system Blockage (RAS), calcium channel blocker and combined drugs on TWEAK, PTX3 and FMD levels in Diabetic Proteinuric Patients with Hypertension' (ClinicalTrials.gov Identifier:NCT00921570). The investigators will use the samples of the some patients for this study. The investigators also registered the study 'FGF-23 and Endothelial Dysfunction in Diabetic Proteinuric Patients' (ClinicalTrials.gov Identifier: NCT01703234). The investigators will combine these two registered studies (NCT00921570 and NCT01703234) in one study.

DETAILED DESCRIPTION:
The patients who were non-obese (BMI<30kg/m2), non dyslipidemic (total cholesterol <200mg/dl, Triglyceride<150mg/dl), and free of cardiovascular events (negative medical history, negative ECG findings) were investigated for enrollment. CKD stage 1 patients older than 18 years of age and willing to participate to the study were screened. From the 231 patients with established type 2 diabetes mellitus, 126 had proteinuria and/or hypertension (24 h protein excretion 1-2 g/day, systolic blood pressures ≥140mmHg and/or diastolic blood pressures ≥ 90 mmHg, respectively). All cases were first referrals and at the time of the study all were off treatment. Patients with history of coronary artery disease, smokers and those taking statins or renin-angiotensin blockers were excluded because of the effect of these factors on endothelial dysfunction. Of 61 screened patients 32 met the study criteria and were included in this study. The duration of proteinuria and diabetic nephropathy after initial diagnosis was not known.

The exclusion criteria were as follows: A)Nephrotic syndrome, B)coronary heart disease (patients with ischemic ST-T alterations and voltage criteria for LVH on electrocardiogram, and with history of revascularization or myocardial infarction), C) elevated liver enzymes (AST or ALT levels ≥ 40U/L) and D) renal failure (serum creatinine levels > 1.3 mg/dl). In order to evaluate the effect of calcium channel blocker on serum FGF-23 concentrations, patients with proteinuria were given an calcium channel blocker (Amlodipine 10 mg/day) for 12 weeks. The effect of calcium channel blocker on insulin sensitivity and proteinuria was also investigated.

After the intervention period, blood samples were obtained for assay of plasma PTX3 concentrations, HbA1c , and insulin resistance scores (HOMA-IR).

Urine samples were also collected over a 24-hour period to determine the degree of proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 1 patients
* Older than 18 years of age
* Type 2 Diabetic patients
* Proteinuria

Exclusion Criteria:

* History of coronary artery disease
* Smokers
* Taking statins or renin-angiotensin blockers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Fibroblast Growth factor 23

SECONDARY OUTCOMES:
Flow mediated dilatation

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Yilmaz MI, Sonmez A, Saglam M, Kurt YG, Unal HU, Karaman M, Gok M, Cetinkaya H, Eyileten T, Oguz Y, Vural A, Mallamaci F, Zoccali C. Ramipril lowers plasma FGF-23 in patients with diabetic nephropathy. Am J Nephrol. 2014;40(3):208-14. doi: 10.1159/000366169. Epub 2014 Oct 10. PMID 25324042